CLINICAL TRIAL: NCT03331887
Title: One Year Clinical Evaluation of E-max CAD Crowns Retained With Fiber Reinforced Composite Post Versus E-max CAD Endocrowns in Anterior Endodontically Treated Teeth: A Randomized Clinical Trial
Brief Title: E-max CAD Crowns Retained With Fiber Reinforced Composite Post Versus E-max CAD Endocrowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Hesham Abou El-Enein, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-10-28
Record Dates: First submitted 2017-10-29; First posted 2017-11-06 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Tooth Fractures; Debonding
Keywords: endodontically treate teeth; Emax crowns; Fiber reinforced composite post; Endocrowns
MeSH Terms: conditions — Tooth Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-max CAD crowns retained with Fiber Reinforced Composite Post (Active Comparator): The modulus of elasticity of FRC post is (18-22 GPa) resembling that of dentin. Ideally the remaining tooth, the fiber post and the composite cement create a "monoblock" in which the loads are uniformly dissipated, ensuring a behavior similar to healthy teeth with a lower risk of root fracture. Using lithium disilicate e.max restorations is documented in literature as a successful restoration.
  Interventions: Procedure: E-max CAd crowns retained with fiber reinforced composite post
- E-max CAD Endocrowns (Experimental): Endocrowns have several advantages over conventional crowns like adequate function and esthetic with less chair time reduced number of interfaces in the restorative system. Stress concentration is less because of the reduction in the nonhomogenous material present. The preparation design is conservative compared to the traditional crown. Supragingival margin prevents interferences with periodontal tissues so involvement of the biological width is minimal. The application and polymerization of resins is also better controlled. Emax ceramic material have a high mechanical strength and are capable of being acid etched, with the adhesive capacity of adhesive systems and resinous cements, made it possible to restore endodontically treated teeth, without cores and intraradicular posts.
  Interventions: Procedure: E-max CAD endocrown

INTERVENTIONS:
Procedure: E-max CAD endocrown — endocrown used to restore endodontically treated teeth with E-max CAD endocrowns
  Arms: E-max CAD Endocrowns
Procedure: E-max CAd crowns retained with fiber reinforced composite post — fiber reinforced composite post need to restore endodontically treated tooth with E-max crown
  Arms: E-max CAD crowns retained with Fiber Reinforced Composite Post

SUMMARY:
Different types of post and core have been used for several years for restoring anterior endodontically treated teeth, but their preparations involve various risks such as: root perforation, root weakness and tooth fracture. The introduction of adhesive systems and conservative restorations, make it possible to reconstruct damaged anterior endodontically treated teeth with conservative restoration as endocrowns. The hypothesis of this trial is that E-max CAD endocrowns will show comparably equal clinical performance if compared to E-max CAD crowns retained with fiber reinforced composite post and core system when treating anterior endodontically treated teeth..

DETAILED DESCRIPTION:
This trial will be conducted on patients from the out patient clinic in the fixed prosthodontics clinic, Faculty of Oral and Dental Medicine, Cairo University.

* Adherence session will take place in the presence of the patients in the initial visit. This include that the patients will be informed by Abou El-Enein Y about the study steps and maintenance of oral hygiene instructions. Participant will be asked by Abou El-Enein Y if they have any problem like pain.
* Motivation and enforcing the maintenance of oral hygiene measures by Abou El-Enein Y.

The visits will be designed as follow:

* st visit: (Y.A) will call participants before tooth preparation procedure for preoperative records, face to face adherence reminder session, clinical examination, radiograohic examination, pre-operative photographing, Impression taking for study cast analysis and waxing up. Each participant will be asked to sign consent form written in patient native language.

  2nd visit: Tooth preparation for either e-max crown retained with fiber reinforced composie post or e-max endocrown, secondary impression and temporarization.

  3rd visit: Try in of the restoration.

  4th visit: Participants will be called again for final cementation.

  5th visit: Follow up.

Sample size: 12 in each group to be able to reject the null hypothesis that the rates for case and controls are equal with probability (power) 0.8. This number is to be increased to 16 in each group to compensate for possible losses during follow up.

Recruitment: The patients fulfill inclusion criteria will be selected from dental clinics of the Fixed Prosthodontics Department - Cairo University (internal recruitment).

Screening of patients will carried out until target number is reached (consecutive sampling).

Methods: Assignment of interventions:

Sequence generation: Radi I (R.I) will allocate participants in two different groups with 1:1 allocation ratio by using computerized sequence generation (www.randomizer.org).

Implementation: IR will be responsible for provide allocation generation and save it in the envelopes in secured place until the date of performing procedure.

Plans to promote participant retention & complete follow up: Telephone numbers of each patients and address will be taken and included in study, then phone calls and messages will be sent to remind patients before each appointment.

Data management: Guindy J (G.J) will enter all data electronically. Patient files are to stored in numerical order in a secured place in locked cabinets. G.J and Z.A will have access to data . Categorical data will be described as numbers and percentages. Data will be explored for normality using Kolmogrov-Smirnov test and Shapiro-Wilk test. Comparisons between two groups for normally distributed numeric variables will be done using the Student's t-test while for non normally distributed numeric variables will be done by Mann-Whitney test. Comparisons between categorical variables will be performed using the chi square test. A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed. Statistical Methods will be done using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 21 (SPSS Inc., Chicago, IL).

Data Monitoring: Z.A will be responsible of data monitoring if any lost or delete occurs, in that case: back up data will be taken from (G.J) to provide hard copy for the requested data for Z.A.

Harms: If 50% of the patients showed any unfavorable signs as sever pain, irreparable fracture or shade changes which might affect the results. Then the treatment will be considered as stopped guidelines which necessitate stopping the treatment and interim analysis will be performed.

Consent: Researcher will discuss the trial with all patients. Then patient can have an informed discussion with the researcher. Researcher will obtain written consent from patients willing to participate in the trial. All consent forms will write in Arabic language (Appendix 1.1).

Access to data: The supervisors (Z.A and G.J) will give access to the data sets. All data sets will be protected by password. To ensure confidentiality, Participant study information will become confidentially.

Ancillary and post-trial care: All patients will be followed up 2 years even after the trial ends to report success of the treatments.

Dissemination policy: Study results will be published as partial fulfillment the Requirements for PHD degree in fixed prosthodontics.Topics suggested for presentation or publication will be circulated to the authors.

Data collection: The following assessment surveys (clinical evaluations) will done for both groups: All patients will be recalled after 3, 6, 9, and 12 months. For each recall examination, evaluator will performed the direct clinical evaluation using modified USPHS criteria for margin integrity and gross fracture. In addition, questionnaires will be used to evaluate patients' satisfaction and potential postoperative discomfort

ELIGIBILITY:
Inclusion Criteria:

1. Age range of the patients from 20-60 years old who can read and sign informed consent document. Illiterate patients will be excluded.
2. Patients willing to return for follow-up examinations and evaluation.
3. Medically free patients or with controlled systemic disease.
4. No active periodontal disease.
5. Patients with anterior endodontically treated tooth/teeth indicated for Endocrown restoration (e.g. teeth without missing any wall, 2-3mm of sound tooth structure above cement-enamel junction).

Exclusion Criteria:

1. Patients under 20 years old.
2. Patients with bad oral hygiene and motivation.
3. Patients with psychiatric problems or unrealistic expectation (patient have phobia from dental treatments or needle bricks).
4. Patients with missing teeth opposing to the area intended for restoration.
5. Patients with parafunctional habits (clencing /bruxism).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Gross Fracture | 12 months
  it indicates if the restoration is intact and fully retained or not using USPHS criteria for recording Categorical Alpha (A):Restoration is intact and fully retained.Bravo (B):Restoration is partially retained with some portion of the restoration still intact.Charlie (C):Restoration is completely missing

SECONDARY OUTCOMES:
Patient Satisfaction | 12 months
  measured using Visual Analogue scale For Endocrowns:Are you satisfied with your endocrown appearance? Are you satisfied with your endocrown shade Do you feel your endocrown are poorly aligned? Do you feel your endocrown are protruding?Are you hiding your teeth while smiling? For E-max crowns retained with fiber reinforced composite post: Are you satisfied with your crown appearance? Are you satisfied with your crown shade?Do you feel your crown are poorly aligned? Do you feel your crown are protruding?Are you hiding your teeth while smiling
Marginal Integrity | 12 months
  Alpha (A):The explorer does not catch and no visible crevice along the periphery of the restoration.Bravo (B):The explorer catches and there is visible evidence of a crevice, which the explorer penetrates, indicating that the edge of the restoration does not adapt closely to the tooth structure. The dentin and/or the base is not exposed, and the restoration is not mobile.Charlie ©: The explorer penetrates and extended to the dento-enamel junction.

IPD SHARING:
Plan to Share IPD: No